CLINICAL TRIAL: NCT04123171
Title: Cerebrovascular Correlates of Dementia in Community-dwelling Older Adults Living in Remote Rural Communities - The Three Villages Study. Methodology and Operational Definitions.
Brief Title: Cerebrovascular Correlates of Dementia in Rural Communities - The Three Villages Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Oscar H. Del Brutto, Researcher, Universidad de Especialidades Espiritu Santo
Other Study IDs: 201901UEES
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Dementia; Cardiovascular Risk Factor; Atherosclerosis; Cerebral Small Vessel Diseases; Cognitive Decline
Keywords: Dementia; Cognitive performance; Vascular diseases; Rural Ecuador; Atahualpa; El Tambo; Prosperidad; Three villages study
MeSH Terms: conditions — Dementia; Atherosclerosis; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Three Villages Cohort: Individuals aged 60 years or more identified by means of door-to-door surveys, living in Atahualpa, El Tambo, and Prosperidad. Individuals will be interviewed with validated field instruments, and there will be invited for the practice of complementary exams to recognize markers of aterosclerosis and cerebral small vessel disease.
  Interventions: Diagnostic Test: Neuroimaging studies

INTERVENTIONS:
Diagnostic Test: Neuroimaging studies — Complementary exams are not invasive and will be performed in enrolled individuals who sign a comprehensive informed consent form
  Other Names: Ultrasound examinations; Ankle-brachial index determinations

SUMMARY:
This study aims to assess the prevalence and severity of dementia in an established cohort of community-dwelling older adults living in three neighboring rural Ecuadorian villages (Atahualpa, El Tambo, and Prosperidad), as well as to evaluate clinical and neuroimaging correlates of dementia in the study population. By the use of the Clinical Dementia Rating Scale (CDRS), the study also aims to assess the lower cutoff of the MoCA that better correlates with the occurrence of dementia in the study population. In addition, this study will provides grounds for the initiation of a prospective cohort study to assess factors influencing the development of dementia in the follow-up.

DETAILED DESCRIPTION:
The Three Villages Study is a population-based prospective cohort study designed to reduce the increasing burden of cognitive decline and dementia in rural Ecuador. Before the study, our Executive Committee met with community leaders to explain the aims of the study and to learn about the culture and traditions of villagers. Field personnel were trained to assure uniformity in data collection. With the aid of satellite view (Google Earth, Google Inc., Mountain View, CA), updated sketches of the villages were performed to identify blocks and houses.

The study initially will follow a 3-Phase cross-sectional design. During Phase I, Atahualpa, El Tambo, and Prosperidad residents aged 60 years or more will be identified by means of a door-to-door survey and interviewed with validated questionnaires to identify those with relevant risk factors and suspected conditions of interest. In Phase II, certified neurologists will examine suspected cases as well as random samples of negative individuals, to assess reliability of field instruments and to determine prevalence of the investigated conditions. In Phase III, enrolled individuals will be invited to undergo complementary tests. Thereafter, incoming residents will be recruited and followed-up by means of yearly door-to-door surveys and other overlapping sources to estimate incidence of the disorders of interest.

ELIGIBILITY:
Inclusion Criteria: Individuals aged 60 years of more residing in Atahualpa, El Tambo, and Prosperidad, who signed a comprehensive informed consent form.

-

Exclusion Criteria: Severely disabled individuals in whom interviews and procedures cannot be performed

-

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Atahualpa, el Tambo and Prosperidad are representative of rural villages of Coastal Ecuador, and were selected because they achieve several requisites to be considered optimal settings for the practice of epidemiological studies. The villages have a low index of migration rate. Inhabitants are homogeneous regarding race/ethnicity, lifestyles and diet, which is rich in oily fish. Residents are Ecuadorian natives with little evidence of cross-breading (Amerindians). Almost all men belong to the blue-collar class and most women are homemakers.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence and severity of dementia in the study population | One year
  The Clinical Dementia Rating Scale will be applied to all participants
To assess cerebrovascular correlates of mild cognitive impairment and dementia in the study population | One year
  Neuroimaging studies, ultrasound examination of extracranial carotid arteries, and ankle-brachial index determinations will be used to assess the presence of large vessel aterosclerosis and cerebral small vessel disease in the study population
To assess cognitive decline in the follow-up | five years
  Enrolled individuals will be prospectively followed every year for up to five years, and will be re-assessed to determine the progression of cognitive impairment and its relationship with markers of aterosclerosis and cerebral small vessel disease

SECONDARY OUTCOMES:
To assess cutoffs of the Montreal Cognitive Assessment useful to differentiate normal cognitivion from mild cognitive impairment, and mild cognitive impairment to dementia in the study population | five years
  The MoCA was mainly designed to separate normal individuals to those with MCI. However, a major limitation of the MoCA is its lack of accuracy for identifying persons with dementia. Therefore, the use of more complex field instruments (yet, feasible to apply in individuals living in rural settings) is needed to determine the burden of dementia and its cerebrovascular correlates in rural communities. In this regard, the Clinical Dementia Rating Scale (CDRS) is a useful tool to assess people living in these settings for establishing the burden and severity of dementia as well as to further assess clinical and neuroimaging correlates of this condition.

CONTACTS AND LOCATIONS:
Locations (2):
- Ecuador (2):
  - Universidad de Especialidades Espiritu Santo, Samborondón, Guayas
  - Community Center, Atahualpa, Santa Elena

IPD SHARING:
Plan to Share IPD: Yes
Dta will be available after reasonable request from an investigator for a similar study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2020
Access Criteria: email to the principal investigator

REFERENCES:
- [Result] Del Brutto OH, Penaherrera E, Ochoa E, Santamaria M, Zambrano M, Del Brutto VJ; Atahualpa Project Investigators. Door-to-door survey of cardiovascular health, stroke, and ischemic heart disease in rural coastal Ecuador--the Atahualpa Project: methodology and operational definitions. Int J Stroke. 2014 Apr;9(3):367-71. doi: 10.1111/ijs.12030. Epub 2013 Mar 19. PMID 23506643
- [Result] Del Brutto OH, Mera RM, Peralta LD, Hill JP, Generale LM, Torpey AP, Sedler MJ. Cardiovascular Health Status Among Community-Dwelling Ecuadorian Natives Living in Neighboring Rural Communities: The Three Villages Study. J Community Health. 2020 Feb;45(1):154-160. doi: 10.1007/s10900-019-00728-4. PMID 31446542
- [Result] Del Brutto VJ, Ortiz JG, Del Brutto OH, Mera RM, Zambrano M, Biller J. Total cerebral small vessel disease score and cognitive performance in community-dwelling older adults. Results from the Atahualpa Project. Int J Geriatr Psychiatry. 2018 Feb;33(2):325-331. doi: 10.1002/gps.4747. Epub 2017 May 26. PMID 28548298
- [Result] Del Brutto OH, Mera RM, Del Brutto VJ, Sedler MJ. The bicaudate index inversely associates with performance in the Montreal Cognitive Assessment (MoCA) in older adults living in rural Ecuador. The Atahualpa project. Int J Geriatr Psychiatry. 2016 Aug;31(8):944-50. doi: 10.1002/gps.4419. Epub 2016 Feb 2. PMID 26833914
- [Result] Del Brutto OH, Mera RM, Castillo PR, Del Brutto VJ. Key findings from the Atahualpa Project: what should we learn? Expert Rev Neurother. 2018 Jan;18(1):5-8. doi: 10.1080/14737175.2018.1400382. Epub 2017 Nov 6. No abstract available. PMID 29088979